CLINICAL TRIAL: NCT06284122
Title: A Phase III Randomized, Open-label, International, Multicenter Study Evaluating the Efficacy and Safety of Mosunetuzumab Plus Lenalidomide in Comparison to Anti-CD20 Monoclonal Antibody Plus Chemotherapy in Subjects With Previously Untreated FLIPI 2-5 Follicular Lymphoma
Brief Title: Study of Mosunetuzumab Plus Lenalidomide Compared to Anti-CD20 Anti-body + Chemotherapy in Follicular Lymphoma FLIPI2-5
Acronym: MorningLyte
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Lymphoma Study Association (Other); Swiss Cancer Institute (Other); Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MorningLyte
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Lenalidomide; Rituximab; obinutuzumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Mosun-Len (Experimental): Mosunetuzumab + lenalidomide
  Interventions: Drug: Mosunetuzumab; Drug: Lenalidomide
- R-CHOP (Active Comparator): Rituximab-CHOP
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristin; Drug: Prednisone
- G-CHOP (Active Comparator): Obinutuzumab-CHOP
  Interventions: Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristin; Drug: Prednisone
- R-Benda (Active Comparator): Rituximab-Bendamustin
  Interventions: Drug: Rituximab; Drug: Bendamustin
- G-Benda (Active Comparator): Obinutuzumab-Bendamustin
  Interventions: Drug: Obinutuzumab; Drug: Bendamustin

INTERVENTIONS:
Drug: Mosunetuzumab — 5 mg (step-up dosing) Day 1 of C1 45 mg Day 8 and Day 15 of C1, 45 mg Day 1 from C2 to C12, 45 mg Day 1 from C13 to C21
  Arms: Mosun-Len
Drug: Lenalidomide — 20 mg/day Day 1 to Day 21 from C2 to C12
  Arms: Mosun-Len
Drug: Rituximab — when associated to CHOP IV 375mg/m² SC 1400 mg allowed from C2 Day 1 of C1 Day 1 from C2 to C6 Day 1 from C7 to C20
  Arms: R-CHOP
Drug: Obinutuzumab — when associated to CHOP 1000 mg Day 1, Day 8, Day 15 of C1 Day 1 from C2 to C8 Day 1 from C9 to C18
  Arms: G-CHOP
Drug: Cyclophosphamide — 750 mg/m2 Day 1 from C1 to C6
  Arms: G-CHOP; R-CHOP
Drug: Doxorubicin — 50 mg/m2 Day 1 from C1 to C6
  Arms: G-CHOP; R-CHOP
Drug: Vincristin — 1.4 mg/m2 (cap cf. below)$ Day 1 from C1 to C6
  Arms: G-CHOP; R-CHOP
Drug: Prednisone — 100 mg/day Day 1 to Day 5 from C1 to C6
  Arms: G-CHOP; R-CHOP
Drug: Rituximab — when associated to bendamustin IV 375mg/m² SC 1400 mg allowed from C2 Day 1 of C1 Day 1 from C2 to C6 Day 1 from C7 to C18
  Arms: R-Benda
Drug: Obinutuzumab — when associated to bendamustin 1000 mg Day 1, Day 8, Day 15 of C1 Day 1 from C2 to C8 Day 1 from C9 to C20
  Arms: G-Benda
Drug: Bendamustin — 90 mg/m2 Day 1 and Day 2 from C1 to C6
  Arms: G-Benda; R-Benda

SUMMARY:
This study is a phase III, randomized, open-label, international, multicenter, interventional trial, designed to compare the efficacy and safety of mosunetuzumab in combination with lenalidomide versus anti-CD20 monoclonal antibody (mAb) plus chemotherapy in patients with previously untreated FLIPI 2-5 follicular lymphoma.

DETAILED DESCRIPTION:
This study is a phase III, randomized, open-label, international, multicenter, interventional trial, designed to compare the efficacy and safety of mosunetuzumab in combination with lenalidomide versus anti-CD20 monoclonal antibody (mAb) plus chemotherapy in patients with previously untreated Follicular Lymphoma International Prognostic Index (FLIPI) 2-5 follicular lymphoma This study is composed of a screening period (up to 6 weeks before randomization, i.e., 42 days), a treatment period (30 months i.e., 125w), a safety follow-up period (90 days i.e., 3 months), and a survival follow-up period (up to 7 years after the last randomized patient). The enrollment will last approximately 34 months. The total duration of the study will be therefore approximately 10 years.

Once a patient provides written consent, they may enter the screening phase, with a duration up to 6 weeks prior to randomization and initiation of treatment.

Upon completion of the required assessments in the screening phase, and fulfillment of the eligibility criteria, patients will be randomized. Investigators will be requested to indicate their treatment choice among permitted immuno-chemotherapy regimens just before randomization.

The treatment period for each patient starts with the first intake. The patients will receive protocol-specified treatments until:

* inability to achieve a response at the end of induction phase (at M12 evaluation for experimental arm, and at M6 evaluation for control arms),
* relapse or progression of the disease,
* withdrawal of consent,
* or unacceptable toxicity

In the experimental arm, patients will be treated for 1 cycle of 3 weeks for mosunetuzumab and then 11 cycles of 4 weeks for mosunetuzumab and lenalidomide (47 weeks, around 11 months) during the induction phase, and for a maximum of 9 additional cycles of 8 weeks during the maintenance phase (72 weeks, around 17 months), up to around 125 weeks (30 months). Patients should start the maintenance phase 7 to 8 weeks after the start of last induction cycle (C12).

In the control arm, patients will be treated for 8 or 6 cycles of 3 or 4 weeks for anti-CD20 mAb +cyclophosphamide-doxorubicine-vincristine-prednisone (CHOP) or anti-CD20 mAb + Bendamustine, respectively, depending on the assigned arm (24 weeks, around 5 months) during the induction phase, and for a maximum of 12 additional cycles of 8 weeks during the maintenance phase (96 weeks, around 22 months), up to around 125 weeks (30 months). Patients should start the maintenance phase, 6 to 7 or 7 to 8 weeks after the start of last induction cycle (C8 or C6).

The option to cross-over from the control arm to the experimental arm is not allowed.

All randomized patients will be followed for progression-free survival and overall survival using the same schedule. Patients will be followed up from End of treatment evaluation every 3 months during the first two years, then every 6 months during the next 3 years, then yearly until the end of study.

The end of study will occur when all randomized patients have been followed-up for survival for at least 7 years (or discontinued study early).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically proven previously untreated CD20+ follicular lymphoma grade 1, 2, or 3a (including patient watched during up to 10 years after initial diagnosis) as assessed by the investigators according to the World Health Organization (WHO) 2016 classification12, or classical follicular lymphoma according to the WHO 2022 classification13. Diagnostic tissue must be available for central pathology review, exploratory endpoints and secondary data use. (Patients with absolute lymphocyte count > 20 G/L must be discussed with the Sponsor before screening/inclusion).
2. FLIPI 2-5.
3. All Ann Arbor stages (including stage I if FLIPI ≥ 2).
4. Must need treatment as evidenced by at least one of the following criteria:

   * Bulky disease defined as:
   * a nodal or extranodal mass/lesion > 7 cm in its largest diameter or,
   * involvement of at least 3 nodal or extranodal sites (each with a diameter greater than > 3 cm)
   * Presence of at least one of the following B symptoms:
   * fever (> 38°C) of unclear etiology
   * night sweats
   * weight loss greater than 10% within the prior 6 months
   * Symptomatic splenomegaly
   * Any compressive syndrome (for example, but not restricted to- ureteral, orbital, gastrointestinal)
   * Any one of the following cytopenias due to lymphoma:
   * hemoglobin < 10g/dL (6.25 mmol/L)
   * platelets <100 x 109/L, or
   * absolute neutrophil count (ANC) < 1.5 x 109/L
   * Pleural or peritoneal serous effusion (irrespective of cell content)
   * β2microglobulin > ULN or lactate dehydrogenase (LDH) > ULN
5. At least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extra nodal lesion, defined as > 1.0 cm in its longest dimension (and 18F-2-fluoro-2-deoxy-D-glucose (FDG)-avid lesion).
6. Patient who understood and voluntarily signed and dated an informed consent prior to any study-specific assessments/procedures.
7. Must be ≥ 18 years at the time of signing the informed consent form (ICF).
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
9. Estimated minimum life expectancy of 3 months.
10. Adequate hematological function within 28 days prior to signing informed consent, including:

    * Absolute neutrophil count (ANC) ≥ 1 x 109/L
    * Platelet count ≥ 75 x 109/L, or ≥ 30 x 109/L if bone marrow infiltration or splenomegaly
    * Hemoglobin ≥ 8.0 g/dL (5 mmol/L) unless related to bone marrow infiltration or splenomegaly. Transfusion is allowed before starting treatment (no required window)
11. Normal laboratory values:

    * Measured or estimated creatinine clearance ≥ 40 mL/min calculated by institutional standard method (MDRD or Cockcroft-Gault)
    * aspartate aminotransferase (AST) or alanine aminotransférase (ALT) ≤ 2.5 x the upper limit of normal (ULN), except in patients with documented liver or pancreatic involvement by lymphoma ≤ 5 x ULN
    * Serum total bilirubin ≤ 1.5 x ULN (or ≤ 3 x ULN for patients with Gilbert syndrome), except in patients with documented liver or pancreatic involvement by lymphoma ≤ 3 x ULN
12. left ventricular ejection fraction (LVEF) within normal range (i.e. > 50% as evaluated by Transthoracic Echocardiography or > 45% as evaluated by isotopic method (MUGA scan)).
13. Patients should be able to receive adequate prophylaxis and/or therapy for thromboembolic events (aspirin, low molecular weight heparin or direct oral anticoagulants).

    Patients with a curative anticoagulation therapy can be enrolled. A patient with deep vein thrombosis due to compressive syndrome is eligible if a curative anticoagulation therapy has been started at least 1 week before initiating study treatment: low molecular weight heparin possible at treatment onset, then direct oral anticoagulants according to local practices.
14. Must be able to adhere to the study visit schedule and other protocol requirements.
15. Negative SARS-CoV-2 test within 7 days prior to randomization. Rapid antigen test is also acceptable. If a patient has a positive SARS-CoV-2 test before randomization, another test should be done and be negative within 7 days before initiation of treatment.
16. Negative HIV test before randomization, with the following exception:

    Patients with a positive HIV test before randomization are eligible provided they are stable on antiretroviral therapy for at least 4 weeks, have a CD4 count ≥ 200/ µL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months.
17. For women of childbearing potential (WOCBP) (refer to section 14.7): must have a negative result for pregnancy test (highly sensitive serum) at screening and within 7 days before initiation of study treatment, and agree to abstain from breastfeeding during study participation, and for at least 28 days after the final dose of lenalidomide (if applicable), 3 months after the final dose of mosunetuzumab and tocilizumab (if applicable), 6 months after the final dose of chemotherapies (if applicable), 12 months after the final dose of rituximab (if applicable), and 18 months after the final dose of obinutuzumab (if applicable).
18. For men (refer to section 14.7): Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: with a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period (including periods of treatment interruption), and for at least 28 days after the final dose of lenalidomide (if applicable), 2 months after the final dose of tocilizumab (if applicable), 6 months after the final dose of chemotherapies (if applicable), 12 months after the final dose of rituximab (if applicable), and 3 months after the final dose of obinutuzumab (if applicable).
19. Patient covered by any social security system (France).
20. Patient who understands and speaks one of the country official languages, unless local regulation authorizes independent translators.

Exclusion Criteria:

1. Grade 3b follicular lymphoma according to the WHO 2016 classification12, or follicular large B-cell lymphoma according to the WHO 2022 classification13.
2. Suspicion or clinical evidence of transformed lymphoma at enrollment by investigator assessment (e.g., high SUV in at least one lesion that was not biopsied, and discordant with SUV of biopsied lesion (at least double of the average SUV), LDH > 2.5 x ULN especially in a context of rapidly progressive disease, etc. (Please contact the Sponsor to discuss any possible inclusion in borderline cases or any doubt)
3. Prior localized radiotherapy for the FL.
4. Prior history of another lymphoma.
5. Uncontrolled symptomatic pleural or serous effusion requiring urgent treatment within 48 hours (patients with controlled disease after adequate pleural/serous drainage and/or effective pleurX™ or similar system are eligible).
6. Uncontrolled symptomatic ureterohydronephrosis resulting in renal failure (patients with adequate management i.e. ureteral catheter or double J stent allowing renal failure control are eligible).
7. Symptomatic lymphomatous epidural lesion (patients whose disease is controlled by neurosurgery or short course of steroids are eligible).
8. Use of any standard or experimental anti-cancer drug therapy within 42 days of the start (Day 1) of study treatment.
9. Systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) or corticosteroid > 1mg/kg/day prednisone or equivalent within 10 days prior to first dose of study treatment. Systemic corticosteroid treatment < 20 mg/day of prednisone or equivalent, inhaled corticosteroids and mineralocorticoids for management of orthostatic hypotension is permitted. A single dose of dexamethasone for nausea or B symptoms is permitted.
10. Received a live, attenuated vaccine within 4 weeks before the first dose of study treatment, or in whom it is anticipated that such a live attenuated vaccine will be required during the study period or within 5 months after the final dose of study treatment.
11. Major surgery (excluding surgical documentation of FL) within 28 days prior to signing informed consent.
12. Seropositive for or active viral infection with Hepatitis B virus (HBV):

    * HBsAg positive
    * HBsAg negative, anti-HBs positive and/or anti-HBc positive and detectable viral DNA (Patients who are HBsAg negative, anti-HBs positive and/or anti-HBc positive but viral DNA negative are eligible. They should be treated and perform testing at regular interval; Patients who are seropositive due to a history of hepatitis B vaccine (anti-HBs positive) are eligible).
13. Known seropositive for, or active infection hepatitis C virus (HCV) (Patients who are positive for HCV antibody with a negative viral RNA are eligible).
14. Known or suspected hypersensitivity to biopharmaceuticals produced in Chinese hamster ovarian (CHO) cells or any component of the mosunetuzumab, Anti-CD20 mAb, tocilizumab, lenalidomide formulation, including mannitol; or to any of the excipients.
15. History of solid organ transplantation or allogeneic stem cell transplant (SCT).
16. Active autoimmune disease requiring treatment.
17. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

    * Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
    * Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Participants with a history of disease-related immune thrombocytopenic purpura or autoimmune hemolytic anemia may be eligible.
    * Participants with a remote history of, or well-controlled autoimmune disease, with a treatment-free interval from immunosuppressive therapy for 12 months may be eligible after review and discussion with the Primary investigator.
18. Participants with any active infection such as known active bacterial, viral (including SARS-CoV-2), fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds), known or suspected chronic active Epstein-Barr virus (EBV) infection, are excluded.
19. Evidence of any significant, concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to:

    * significant cardiovascular disease [e.g., Objective Class C or D heart diseases (cf. Classes of Heart Failure | American Heart Association), myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina)
    * significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
    * clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
    * current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 1 year and have no residual neurologic deficits as judged by the investigator are allowed. Participants with a history of epilepsy who have had no seizures in the past 2 years with or without anti-epileptic medications can be eligible.
20. History of confirmed progressive multifocal leukoencephalopathy (PML).
21. Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
22. History of erythema multiforme, Grade ≥3 rash, or blistering rash following prior treatment with immunomodulatory derivatives.
23. History of interstitial lung disease (ILD), drug-induced pneumonitis, and autoimmune pneumonitis.
24. Active malignancy other than the one treated in this research. Prior history of malignancies unless the patient has been free of the disease for ≥ 3 years. However, patients with the following history/concurrent conditions are eligible:

    * Localized non-melanoma skin cancer.
    * Carcinoma in situ of the cervix.
    * Carcinoma in situ of the breast.
    * Incidental histologic finding of prostate cancer (T1a or T1b as per Tumor Node Metastasis (TNM) staging system) or prostate cancer that has been treated with curative intent.
25. Presence or history of CNS or meningeal involvement by lymphoma.
26. Pregnant, planning to become pregnant or lactating WOCBP.
27. Any significant medical conditions, including the presence of laboratory abnormality or psychiatric illness which places the patient at unacceptable risk if he/she were to participate in the study, and likely to interfere with participation in this clinical study (according to the investigator's decision) or which confounds the ability to interpret data from the study.
28. Person deprived of his/her liberty by a judicial or administrative decision.
29. Person hospitalized without consent.
30. Adult person under legal protection.

Nota bene: for 28., if there is an individual benefit for such patients, an Ethics Committee will have to be informed case by case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 130 PFS events assessed by an Independent Review Committee (IRC) (4.6 years)
  time from randomization to the date of first documented disease progression/relapse or death from any cause, by Lugano 2014
Progression Free Survival (PFS) | 173 PFS events assessed by IRC (5.8 y)
  time from randomization to the date of first documented disease progression/relapse or death from any cause, by Lugano 2014

SECONDARY OUTCOMES:
Overall Response (OR) | 6 months
  by Lugano 2014, assessed by investigator and IRC
Complete Metabolic Rate (CMR) | 6 months
  by Lugano 2014, assessed by investigator and IRC
Overall Response (OR) | 12 months
  by Lugano 2014, assessed by investigator and IRC
Complete Metabolic Rate (CMR) | 12 months
  by Lugano 2014, assessed by investigator and IRC
Best Overall Response (CMR + PMR) rate | 4.6 years
  by Lugano 2014, assessed by investigator and IRC
Best Overall Response (CMR + PMR) rate | 5.8 years
  by Lugano 2014, assessed by investigator and IRC
Progression of disease within 2 years (POD24) | 2 years
  rate of progression of disease (POD) within 2 years of first line therapy
PFS | 4.6 years
  by Lugano 2014, assessed by investigator
PFS | 5.8 years
  by Lugano 2014, assessed by investigator
Event Free Survival (EFS) by Lugano 2014 | 4.6 years
  time between randomization and date of first documented disease progression/relapse, initiation of a new anti-lymphoma treatment or death from any cause
Event Free Survival (EFS) by Lugano 2014 | 5.8 years
  time between randomization and date of first documented disease progression/relapse, initiation of a new anti-lymphoma treatment or death from any cause
Time to Next Anti-Lymphoma Treatment (TTNLT) | 4.6 years
  time between randomization and date of first documented administration of any new anti-lymphoma treatment
Time to Next Anti-Lymphoma Treatment (TTNLT) | 5.8 years
  time between randomization and date of first documented administration of any new anti-lymphoma treatment
Duration of response | 4.6 years
  defined for patients with a best overall response of CMR or PMR determined by Lugano 2014, defined as the time of 1st occurrence of CMR or PMR to disease progression/relapse or death from any cause
Duration of response | 5.8 years
  defined for patients with a best overall response of CMR or PMR determined by Lugano 2014, defined as the time of 1st occurrence of CMR or PMR to disease progression/relapse or death from any cause
Overall Response (OR) | End of treatment (12 months for experimental arm, 6 months for comparative arms)
  assessed by investigator and IRC
Complete Metabolic Rate (CMR) | End of treatment (12 months for experimental arm, 6 months for comparative arms)
  assessed by investigator and IRC
Duration of complete response | 4.6 years
  for patients with a best overall response of CMR determined by Lugano 2014, define as the time of first occurrence of CMR to disease progression/relapse or death from any cause
Duration of complete response | 5.8 years
  for patients with a best overall response of CMR determined by Lugano 2014, define as the time of first occurrence of CMR to disease progression/relapse or death from any cause
Overall Survival (OS) | 4.6 years
  time from randomization to death from any cause
Overall Survival (OS) | 5.8 years
  time from randomization to death from any cause
Incidence and severity of Adverse Events (AE) including Serious and Special Interest AE (SAEs and AESIs) | 4.6 years
Incidence and severity of AEs including SAEs and AESIs | 5.8 years
Tolerability, as assessed by incidence of dose interruptions, delays, dose reductions, and study treatment discontinuation | 4.6 years
Tolerability, as assessed by incidence of dose interruptions, delays, dose reductions, and study treatment discontinuation | 5.8 years
Incidence of Second Primary Malignancies (SPM) | 4.6 years
Incidence of Second Primary Malignancies (SPM) | 5.8 years
anti-drug antibodies (ADA) to mosunetuzumab | each cycle, 18 months, 24 months, 30 months
Time to deterioration in physical functioning | baseline, 6 months, 12 months, 18 months, 24 months, 30 months or end of treatment
  EORTC QLQ-C30 quality of life questionnaire
Time to deterioration in lymphoma symptoms | baseline, 6 months, 12 months, 18 months, 24 months, 30 months or end of treatment
  FACTLym LYMS quality of life questionnaire
Maximum serum concentration of mosunetuzumab - Cmax | each cycle, 18 months, 24 months, 30 months
Minimum serum concentration of mosunetuzumab - Cmin | each cycle, 18 months, 24 months, 30 months
Area under the curve of serum concentration of mosunetuzumab - AUC | each cycle, 18 months, 24 months, 30 months
Maximum serum concentration of lenalidomide - Cmax | each cycle, 18 months, 24 months, 30 months
Minimum serum concentration of lenalidomide - Cmin | each cycle, 18 months, 24 months, 30 months
Area under the curve of serum concentration of lenalidomide - AUC | each cycle, 18 months, 24 months, 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Franck MORSCHHAUSER, Principal Investigator — Lymphoma Study Association; Christian BUSKE, Principal Investigator — GLA
Locations (49):
- Belgium (8):
  - AZ SINT-JAN BRUGGE - OOSTENDE AV - Service Hématologie, Bruges
  - INSTITUT JULES BORDET - Service Hématologie, Brussels
  - UNIVERSITE CATHOLIQUE DE LOUVAIN SAINT-LUC - Service Hématologie, Brussels
  - GRAND HOPITAL DE CHARLEROI - Service Hématologie, Charleroi
  - UNIVERSITAIR ZIEKENHUIS GENT - Service Hématologie, Ghent
  - CHU DE LIEGE - Service Hématologie, Liège
  - CHR VERVIERS - LA TOURELLE - Service Hématologie, Verviers
  - CHU UCL NAMUR - SITE GODINNE - Service Hématologie, Yvoir
- France (37):
  - CH d'AVIGNON - HOPITAL HENRI DUFFAUT - Service d'Onco-Hématologie, Avignon
  - CH DE LA COTE BASQUE - Service Hématologie, Bayonne
  - CHU JEAN MINJOZ - Service Hématologie, Besançon
  - INSTITUT BERGONIE - Service d'Oncologie Médicale, Bordeaux
  - CENTRE HOSPITALIER JEAN ROUGIER - Service d'Oncologie - Hématologie, Cahors
  - CH METROPOLE SAVOIE - SITE CHAMBERY - Service Hématologie, Chambéry
  - CHU ESTAING - Service Thérapie Cellulaire et Hématologie Clinique, Clermont-Ferrand
  - HOPITAL HENRI MONDOR - Unité Hémopathies Lymphoïdes, Créteil
  - CHU DIJON BOURGOGNE - Service Hématologie Clinique, Dijon
  - CHD DE VENDEE - Service Hématologie, La Roche-sur-Yon
  - CHU DE GRENOBLE - Service Hématologie, La Tronche
  - HOPITAL SAINT VINCENT-DE-PAUL - Service Hématologie, Lille
  - CHRU DE LILLE - HOPITAL CLAUDE HURIEZ - Service Hématologie, Lille
  - CHU DE LIMOGES - HOPITAL DUPUYTREN - Service Hématologie Clinique et Thérapie Cellulaire, Limoges
  - INSTITUT PAOLI CALMETTES - Service Hématologie, Marseille
  - CHU DE MONTPELLIER - Département d'Hématologie Clinique, Montpellier
  - GH REGION MULHOUSE ET SUD ALSACE - HOPITAL EMILE MULLER - Service Hématologie, Mulhouse
  - CHU DE NANTES - Service Hématologie, Nantes
  - CENTRE HOSPITALIER DE NIORT - Médecine interne, Niort
  - HOPITAL SAINT-LOUIS - Service Hématologie, Paris
  - CHU DE BORDEAUX - HOPITAL HAUT-LEVEQUE - CENTRE FRANCOIS MAGENDIE - Service d'Hématologie et Thérapie Cellulaire, Pessac
  - CHU LYON-SUD - Hématologie, Pierre-Bénite
  - CHI POISSY SAINT-GERMAIN-EN-LAYE - Service Hématologie, Poissy
  - CHU DE POITIERS - HOPITAL DE LA MILETRIE - Service d'Oncologie Hématologique et Thérapie Cellulaire, Poitiers
  - CH ANNECY GENEVOIS - SITE D'ANNECY - Service Hématologie, Pringy
  - CHU DE REIMS - HOPITAL ROBERT DEBRE - Service Hématologie, Reims
  - CHU PONTCHAILLOU - Hématologie Clinique, Rennes
  - CENTRE HENRI BECQUEREL - Service Hématologie, Rouen
  - INSTITUT CURIE - SITE SAINT-CLOUD - Service Hématologie, Saint-Cloud
  - Institut de Cancérologie et d'Hématologie Universitaire de Saint-Étienne - Service Hématologie, Saint-Priest-en-Jarez
  - INSTITUT DE CANCEROLOGIE STRASBOURG EUROPE - Unité de Recherche Clinique, Strasbourg
  - IUCT ONCOPOLE - Service Hématologie, Toulouse
  - CHU BRETONNEAU - Service Cancérologie - Hématologie et Thérapie Cellulaire, Tours
  - CH DE VALENCIENNES - HOPITAL JEAN BERNARD - Service Hématologie, Valenciennes
  - CHU BRABOIS - Service Hématologie, Vandœuvre-lès-Nancy
  - CH DE BRETAGNE ATLANTIQUE - HOPITAL CHUBERT - Service Hématologie, Vannes
  - GUSTAVE ROUSSY CANCER CAMPUS GRAND PARIS - Département Médecine Oncologique, Villejuif
- Germany (2):
  - UNIVERSITATSKLINIKUM REGENSBURG - Klinik für Innere Medizin III, Regensburg
  - UNIV KLINIKUM ULM - INNERE MEDIZIN III - Service Hématologie, Ulm
- INSTITUTO PORTUGUES DE ONCOLOGIA DE LISBOA FRANCISCO GENTIL - Departamento Hematologia, Lisbon, Portugal
- HOSPITAL CLINICO SALAMANCA - Servicio de Hematologia, Salamanca, Spain